CLINICAL TRIAL: NCT06128967
Title: An Adaptive, Randomized, doublE-blind, Placebo-controlled, Prospective, Pharmacological interVention Study In Participants With Long COVID-19 Syndrome: REVIVE-TOGETHER Trial
Brief Title: A Multicenter, Adaptive, Randomized, doublE-blinded, Placebo-controlled Study in Participants With Long COVID-19: The REVIVE Trial
Acronym: REVIVE
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cardresearch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TOGETHER_REVIVE
Record Dates: First submitted 2023-11-10; First posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Long COVID-19 Syndrome; Chronic Fatigue Syndrome
Keywords: Long COVID-19 Syndrome; Fluvoxamine; Metformin; Adaptive Trial Design; Randomized Controlled Trial
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Fatigue Syndrome, Chronic | interventions — Fluvoxamine

STUDY DESIGN:
Intervention Model Description: Multicenter, adaptive, randomized, double-blind, placebo-controlled, prospective, pharmacological intervention trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The production of medication bottles is carried out by a pharmaceutical company, which does not have access to members of the research centers. The pills are similar in shape, color, size and weight and are packaged in identical bottles and coded according to each medication arm, this code being inaccessible to the investigator, the sponsor, the medical care provider and the research participant.
  The allocation process follows a random sequential distribution into blocks. The posology of the medications is identical for all arms.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo talc pills of same shape, color, weight dispensed in coded bottles. Each bottle contains 120 pills
  Interventions: Drug: Fluvoxamine Maleate 100 MG; Drug: Metformin Extended Release Oral Tablet
- Fluvoxamine 100 mg (Active Comparator): Fluvoxamine maleate 100 mg pills dispensed in coded bottles. Each bottle contains 120 pills
  Interventions: Drug: Placebo
- Metformin XR 750 mg (Active Comparator): Metformin 750 mg Extended release pills dispensed in coded bottles. Each bottle contains 120 pills
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fluvoxamine Maleate 100 MG — Fluvoxamine Maleate 100 mg each pills
  Arms: Placebo
Drug: Placebo — Placebo talc pills of same shape, color, weight if compared with active comparator
  Arms: Fluvoxamine 100 mg; Metformin XR 750 mg
Drug: Metformin Extended Release Oral Tablet — Metformin Extended release oral tablets of 750 mg each pill
  Arms: Placebo

SUMMARY:
Date of notification letter to the IRB informing start of recruitment activities: October 21, 2023.

Long COVID is a multi-systemic condition comprising often severe and persistent symptoms (longer than 12 weeks) that follow a known episode of COVID-19 and cannot be explained by another medical condition. This condition is observed in up to 15% of all individuals after an acute episode of COVID-19, even in those who had a mild and oligosymptomatic SARS-CoV-2 infection. Around 40% of these patients present symptoms that significantly compromise their daily activities.

There is increasing evidence that LONG COVID is accompanied by dysregulated, persistent and uncontrolled inflammation, often accompanied by the development of an autoreactive immune response, including autoantibodies. Symptoms can last months or years, particularly in cases of chronic fatigue syndrome, with significant proportions of individuals having significant chronic impairment, preventing the performance of work and social activities.

DETAILED DESCRIPTION:
There is currently no approved therapies for Long COVID. Several clinical trials have been developed to address this clinical condition, however the results were based on small-scale pilot studies. We developed this adaptive, large-scale, prospective, double-blind clinical trial to evaluate the effect of chronic immune-inflammatory modulation on persistent Long-COVID symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older at the time of screening.
2. Willing and able to provide written informed consent, or with a legal representative who can provide informed consent (where approved locally and nationally).
3. Previous confirmed case of SARS-CoV-2 infection (e.g., reports having a positive nucleic acid amplification test or a professional-use SARS-CoV-2 rapid antigen diagnostic test or positive self-test).
4. Participants with a clinical picture compatible with LONG COVID according to international definitions: (www.nice.org.uk/guidance/ng188, https://www.who.int/publications/i/item/WHO-2019-nCoV-Post_COVID -19_condition-Clinical_case_definition-2021.1), and fatigue symptoms with an average score of at least 03 on the Fatigue Analog Scale (FSS)
5. Not currently hospitalized or requiring hospitalization, or having been hospitalized in an intensive care center at the time of the COVID-19 episode.
6. Participants with the following vital data:

   1. Heart Rate between 55 and 100 bpm;
   2. Temperature below 38o C;
   3. Oxygen saturation ≥ 95%.
7. Patients of childbearing potential or with partners of childbearing potential must agree to use adequate contraception during the study and up to 90 days of follow-up.
8. The symptoms of fatigue cannot be attributed to any other cause (in the researcher's opinion).
9. Willingness to follow all study procedures.

Exclusion Criteria:

1. Known acute SARS-CoV-2 infection;
2. Inability to understand the content of the Informed Consent Form or to follow the study procedures;
3. Known previous diagnosis of malignant encephalomyelitis/chronic fatigue syndrome, unrelated to SARS-CoV-2 infection;
4. Known pre-existing dysautonomia, unrelated to SARS-CoV-2 infection;
5. Diabetes mellitus (exclusion criteria for the Metformin and Metformin Placebo arm);
6. Known stroke within 3 months prior to screening;
7. Known severe anemia, defined as < 8 g/dl;
8. Body Mass Index (BMI) > 35.
9. Known diagnosis of Lyme disease;
10. Any use of illicit drugs not related to marijuana within 30 days prior to informed consent;
11. Pregnant women or women of childbearing age who do not agree to practice an effective method of contraception within 90 days from the date of signing this consent form;
12. Breastfeeding women;
13. Participants using serotonin reuptake inhibitors (donepezil, fluoxetine, escitalopran, parorexitin);
14. Participants chronically using any of the medications under evaluation (metformin and fluvoxamine);
15. Severe current comorbid psychiatric disorder (e.g., clinical depression, anxiety, sleep disorder, eating disorder, substance abuse), uncontrolled and associated with significant symptoms or requiring the use of a medication contraindicated in this research ;
16. Clinical history of moderate to severe hepatic impairment or liver cirrhosis with Child-Pugh classification C or greater;
17. Clinical history of severe lung disease with significant limitation of activities;
18. Inability of the participant to give consent or adhere to the procedures proposed in the study;
19. Taking medications which are known to cause a known side effect of chronic fatigue;
20. Known hypersensitivity and/or intolerance to Fluvoxamine or Metformin;
21. Any clinical condition which, in the investigator's opinion, may prevent participation in this research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2023-10-18 (Actual); Primary Completion 2024-10-18 (Estimated); Study Completion 2025-05-18 (Estimated)

PRIMARY OUTCOMES:
Improvement on Fatigue Severity Score Scale (FSS) | Day 60 after randomization
  Improvement on Fatigue Severity Score Scale (FSS)

SECONDARY OUTCOMES:
Improvement on Fatigue Severity Score Scale (FSS) | Day 30 after randomization
  Improvement on Fatigue Severity Score Scale (FSS)
Improvement on Fatigue Severity Score Scale (FSS) | Day 30 post Study Drug Termination (Day 90 after randomization)
  Improvement on Fatigue Severity Score Scale (FSS)
Reduction on any cause hospitalization | Day 60 after randomization
  Reduction on any cause hospitalization
Safety of metformin | Since randomization up to Day 60 (last IMP dose)
  Safety of metformin (intention to treat analysis)
Safety of Fluvoxamine | Since randomization up to Day 60 (last IMP dose)
  Safety of Fluvoxamine (intention to treat analysis)
Death of any cause | Since randomization up to Day 60 (last IMP dose)
  Occurrence of Death of any cause

CONTACTS AND LOCATIONS:
Overall Officials: Gilmar Reis, MD,PhD., Study Chair — Cardresearch - Cardiologia Assistencial e de Pesquisa LTDA
Locations (6):
- Brazil (6):
  - CARDRESEARCH - Cardiologia Assistencial e de Pesquisa, Belo Horizonte, Minas Gerais
  - City of Brumadinho, Brumadinho, Minas Gerais
  - Governador Valadares City Public Health Authority, Governador Valadares, Minas Gerais
  - City of Ibirité Public Health Authority, Ibirité, Minas Gerais
  - Sociedade Padrao de Educacao Superior, Montes Claros, Minas Gerais
  - Universidade Federal de Ouro Preto, Ouro Preto, Minas Gerais

IPD SHARING:
Plan to Share IPD: Yes
We are prone to share patient level information data to specific researchers that share the same intention. Data sharing request shall be submitted to a local committee for approval.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: A year after protocol termination
Access Criteria: To be defined